CLINICAL TRIAL: NCT03004859
Title: Eine Beobachtungsstudie Zur Erfassung Von (Asymptomatischem)Vorhofflimmern Mittels Eines Gelegenheitsscreenings älteren Menschen ab 65 Jahren
Brief Title: Opportunistic Screening in Pharmacies for Atrial Fibrillation in Seniors (>65 Years)
Acronym: AF-Stroke
Status: Completed | Type: Observational
Sponsor: RWTH Aachen University (Other)
Collaborators: Apothekerverband Aachen e.V. (Unknown); Pfizer (Industry)
Responsible Party: Principal Investigator, Nikolaus Marx, Univ. Professor Dr. med., RWTH Aachen University
Other Study IDs: 15-073 AF-Stroke
Record Dates: First submitted 2016-11-14; First posted 2016-12-29 (Estimated); Last update posted 2020-03-11 (Actual); Status verified 2018-04

CONDITIONS: Incidence of Atrial Fibrillation in Adults Aged ≥ 65
Keywords: atrial fibrillation; screening; electrocardiogram; community pharmacy; Germany
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Adults ≥ 65 with a positive test result: Adults ≥ 65 that are got a positive test result were asked to visit their general practitioner and are called for an interview two times, 8 weeks and 12 months after the screening in the pharmacy. The results of the data collection and screening in the pharmacies as well as of the two telephone interviews are compared to the results of the adults ≥ 65 with a negative test result.
- Adults ≥ 65 with a negative test result: Adults ≥ 65 that are got a negative test result are called for an interview 12 months after the screening in the pharmacy. The results of the data collection and screening in the pharmacy as well as of the telephone interview are compared to the results of the adults ≥ 65 with a positive test result.

SUMMARY:
Atrial fibrillation (AF) is the most common arrhythmia in Germany and is associated with an increased risk of thromboembolic stroke. The risk to suffer from AF increases with age. Early detection of AF and anticoagulation seem the most effective way of preventing ischaemic stroke in patients at risk. The guidelines of the European Society of Cardiology recommend opportunistic screening for AF by pulse check at each general practitioner visit for all patients aged 65 years or older.

The objective of this study was to test whether an opportunistic AF screening with a hand-held diagnostic tool in a German pharmacy setting is useful in detecting unknown AF among people in the age of 65 and older. Besides a pulse palpation with a hand-held ECG-stick the screening in the pharmacies also includes a questionnaire related to demographics and medical history of the subject as well as several questions concerning the stroke risk stratification (CHA₂DS₂-VASc). Every subject with a positive test result (indication on AF) is insistently asked to make an appointment with his or her general practitioner. The subject receives an information letter for his or her general practitioner that adverts to the positive screening result and the necessity of further diagnostic Investigation.

In order to assess the incidence of unknown AF as well as accomplish the secondary objectives of this study, two follow-ups by means of telephone interviews are performed. First, all subjects with a positive test result are called 8 weeks after the screening in the pharmacies was conducted. The subject is asked several questions concerning personal data/demographics, the stroke risk (CHA₂DS₂-VASc), the medical history regarding to dyspnea and stroke, the bleeding risk (HAS-Bled), the medication, the device, diagnostic, the therapy, the Intervention and the mace. 12 months after the screening in the pharmacies was performed, all participating subjects were called. The list of questions is similar to the one that is used during the first telephone interviews after eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* At least 65 years or older
* Signed informed consent
* Signed subject information

Exclusion Criteria:

* Insufficient language skills
* Limited cognitive abilities
* Limited physical abilities (i.e. tremor)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: All pharmacy customers (male and female) of 65 years and above that meet the inclusion criteria and are not affected by the exclusion criteria are allowed to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 7606 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-08-22 (Actual); Study Completion 2018-08-22 (Actual)

PRIMARY OUTCOMES:
Number of newly detected atrial fibrillation in adults from the age of 65 by means of an opportunistic screening with an ECG hand-held diagnostic tool in a pharmacy setting | 12 months
  The data is going to be collected in a screening period of two weeks in an urban pharmacy setting and a screening period of two weeks of data collection in a more rural pharmacy setting

SECONDARY OUTCOMES:
The subject's behavior change regarding diagnosis and therapy from the ECG measurement at pharmacy at 8 weeks and 12 months. | 8 weeks and 12 Months
  The subject's behavior change is measured by means of a questionnaire, compiled by the research team. The questionnaire is used during the telephone interviews 8 eight weeks and 12 months. The questionnaire includes questions related to personal data/demographics, the stroke risk (CHA₂DS₂-VASc), the medical history regarding to dyspnea and stroke, the bleeding risk (HAS-Bled), the medication, the device, diagnostic, the therapy, the Intervention and the mace.
Identification and description of new therapeutic measures. | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, Professor, Principal Investigator — Head of the Clinic for Cardiology, Pneumology, Angiology and Internal Intensive Medicine
Locations (1):
- Uniklinium RWTH Aachen, Aachen, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] European Heart Rhythm Association; European Association for Cardio-Thoracic Surgery; Camm AJ, Kirchhof P, Lip GY, Schotten U, Savelieva I, Ernst S, Van Gelder IC, Al-Attar N, Hindricks G, Prendergast B, Heidbuchel H, Alfieri O, Angelini A, Atar D, Colonna P, De Caterina R, De Sutter J, Goette A, Gorenek B, Heldal M, Hohloser SH, Kolh P, Le Heuzey JY, Ponikowski P, Rutten FH. Guidelines for the management of atrial fibrillation: the Task Force for the Management of Atrial Fibrillation of the European Society of Cardiology (ESC). Eur Heart J. 2010 Oct;31(19):2369-429. doi: 10.1093/eurheartj/ehq278. Epub 2010 Aug 29. No abstract available. PMID 20802247
- [Background] Chugh SS, Blackshear JL, Shen WK, Hammill SC, Gersh BJ. Epidemiology and natural history of atrial fibrillation: clinical implications. J Am Coll Cardiol. 2001 Feb;37(2):371-8. doi: 10.1016/s0735-1097(00)01107-4. PMID 11216949
- [Background] Heeringa J, van der Kuip DA, Hofman A, Kors JA, van Herpen G, Stricker BH, Stijnen T, Lip GY, Witteman JC. Prevalence, incidence and lifetime risk of atrial fibrillation: the Rotterdam study. Eur Heart J. 2006 Apr;27(8):949-53. doi: 10.1093/eurheartj/ehi825. Epub 2006 Mar 9. PMID 16527828
- [Background] Kaasenbrood F, Hollander M, Rutten FH, Gerhards LJ, Hoes AW, Tieleman RG. Yield of screening for atrial fibrillation in primary care with a hand-held, single-lead electrocardiogram device during influenza vaccination. Europace. 2016 Oct;18(10):1514-1520. doi: 10.1093/europace/euv426. Epub 2016 Feb 6. PMID 26851813
- [Background] Lip GY, Frison L, Halperin JL, Lane DA. Comparative validation of a novel risk score for predicting bleeding risk in anticoagulated patients with atrial fibrillation: the HAS-BLED (Hypertension, Abnormal Renal/Liver Function, Stroke, Bleeding History or Predisposition, Labile INR, Elderly, Drugs/Alcohol Concomitantly) score. J Am Coll Cardiol. 2011 Jan 11;57(2):173-80. doi: 10.1016/j.jacc.2010.09.024. Epub 2010 Nov 24. PMID 21111555
- [Background] Lip GY, Nieuwlaat R, Pisters R, Lane DA, Crijns HJ. Refining clinical risk stratification for predicting stroke and thromboembolism in atrial fibrillation using a novel risk factor-based approach: the euro heart survey on atrial fibrillation. Chest. 2010 Feb;137(2):263-72. doi: 10.1378/chest.09-1584. Epub 2009 Sep 17. PMID 19762550
- [Background] Lloyd-Jones DM, Wang TJ, Leip EP, Larson MG, Levy D, Vasan RS, D'Agostino RB, Massaro JM, Beiser A, Wolf PA, Benjamin EJ. Lifetime risk for development of atrial fibrillation: the Framingham Heart Study. Circulation. 2004 Aug 31;110(9):1042-6. doi: 10.1161/01.CIR.0000140263.20897.42. Epub 2004 Aug 16. PMID 15313941
- [Background] Lowres N, Krass I, Neubeck L, Redfern J, McLachlan AJ, Bennett AA, Freedman SB. Atrial fibrillation screening in pharmacies using an iPhone ECG: a qualitative review of implementation. Int J Clin Pharm. 2015 Dec;37(6):1111-20. doi: 10.1007/s11096-015-0169-1. Epub 2015 Jul 23. PMID 26202627
- [Background] Lowres N, Neubeck L, Redfern J, Freedman SB. Screening to identify unknown atrial fibrillation. A systematic review. Thromb Haemost. 2013 Aug;110(2):213-22. doi: 10.1160/TH13-02-0165. Epub 2013 Apr 18. PMID 23595785
- [Background] Paciaroni M, Agnelli G, Caso V, Venti M, Milia P, Silvestrelli G, Parnetti L, Biagini S. Atrial fibrillation in patients with first-ever stroke: frequency, antithrombotic treatment before the event and effect on clinical outcome. J Thromb Haemost. 2005 Jun;3(6):1218-23. doi: 10.1111/j.1538-7836.2005.01344.x. Epub 2005 May 9. PMID 15892862
- [Background] Pisters R, Lane DA, Nieuwlaat R, de Vos CB, Crijns HJ, Lip GY. A novel user-friendly score (HAS-BLED) to assess 1-year risk of major bleeding in patients with atrial fibrillation: the Euro Heart Survey. Chest. 2010 Nov;138(5):1093-100. doi: 10.1378/chest.10-0134. Epub 2010 Mar 18. PMID 20299623
- [Background] Schnabel RB, Wilde S, Wild PS, Munzel T, Blankenberg S. Atrial fibrillation: its prevalence and risk factor profile in the German general population. Dtsch Arztebl Int. 2012 Apr;109(16):293-9. doi: 10.3238/arztebl.2012.0293. Epub 2012 Apr 20. PMID 22577476
- [Background] Stewart S, Hart CL, Hole DJ, McMurray JJ. A population-based study of the long-term risks associated with atrial fibrillation: 20-year follow-up of the Renfrew/Paisley study. Am J Med. 2002 Oct 1;113(5):359-64. doi: 10.1016/s0002-9343(02)01236-6. PMID 12401529
- [Background] Svennberg E, Engdahl J, Al-Khalili F, Friberg L, Frykman V, Rosenqvist M. Mass Screening for Untreated Atrial Fibrillation: The STROKESTOP Study. Circulation. 2015 Jun 23;131(25):2176-84. doi: 10.1161/CIRCULATIONAHA.114.014343. Epub 2015 Apr 24. PMID 25910800
- [Background] Tieleman RG, Plantinga Y, Rinkes D, Bartels GL, Posma JL, Cator R, Hofman C, Houben RP. Validation and clinical use of a novel diagnostic device for screening of atrial fibrillation. Europace. 2014 Sep;16(9):1291-5. doi: 10.1093/europace/euu057. Epub 2014 May 13. PMID 24825766
- [Background] Vaes B, Stalpaert S, Tavernier K, Thaels B, Lapeire D, Mullens W, Degryse J. The diagnostic accuracy of the MyDiagnostick to detect atrial fibrillation in primary care. BMC Fam Pract. 2014 Jun 9;15:113. doi: 10.1186/1471-2296-15-113. PMID 24913608
- [Background] Wolf PA, Abbott RD, Kannel WB. Atrial fibrillation as an independent risk factor for stroke: the Framingham Study. Stroke. 1991 Aug;22(8):983-8. doi: 10.1161/01.str.22.8.983. PMID 1866765
- [Derived] Zink MD, Mischke KG, Keszei AP, Rummey C, Freedman B, Neumann G, Tolksdorf A, Frank F, Wienstroer J, Kuth N, Schulz JB, Marx N. Screen-detected atrial fibrillation predicts mortality in elderly subjects. Europace. 2021 Jan 27;23(1):29-38. doi: 10.1093/europace/euaa190. PMID 33020819